CLINICAL TRIAL: NCT06894732
Title: To Study the Safety and Efficacy of Disposable Cyclone Ring in Artificial Abortion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChiCTR2400089857
Record Dates: First submitted 2025-01-25; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Induced Abortion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rotary induced abortion (Experimental)
  Interventions: Procedure: Rotary induced abortion

INTERVENTIONS:
Procedure: Rotary induced abortion — Rotary induced abortion under ultrasonic monitoring was performed with intravenous anesthesia.

SUMMARY:
The purpose of this study is to compare the two surgical methods of surgical rotation abortion and surgical negative pressure uterine aspiration with the termination of pregnancy. which one can better protect female fertility; To understand the impact of both surgical approaches on the long-term prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: 20-40 years old, planning to terminate pregnancy; 2) Menopause time≤ 56 days (8 weeks); 3) Ultrasound examination showed early pregnancy in utero, and the average diameter of the fetal sac was 1-3cm; 4) According to the requirements of clinical operation standards, the preoperative examination, laboratory results and surgical indicators are normal 5) The subject was conscious, had good compliance, agreed to participate in the trial, and voluntarily signed the informed consent form

Exclusion Criteria:

* 1) According to the requirements of clinical practice, there are contraindications to induced abortion; 2) The number of previous induced abortions ≥2 times; 3) Diseases affecting uterine cavity morphology such as uterine malformations and uterine fibroids; 4) History of uterine surgery: such as submucosal myomectomy history, mediastinal resection history, uterine adhesion-separation history; 5) Unable to sign the informed consent; 6) Other conditions that the investigator considers inappropriate to participate in this clinical study.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 332 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cervical dilation rate (e.g. %) | 30

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided